CLINICAL TRIAL: NCT03313869
Title: Effects of a Cocktail XXS-2A/Omega-3 on Insulin Sensitivity and Oxidative Stress During a 20-day Period of Physical Inactivity: a Controlled, Randomized Pilot Study on 20 Healthy Men
Brief Title: A Nutrient Cocktail to Protect Against Physical Inactivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre National d'Etudes Spatiales (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CNES
Record Dates: First submitted 2017-10-07; First posted 2017-10-18 (Actual); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Metabolic Disturbance; Glucose Intolerance; Physical Inactivity; Glucose Metabolism Disorders; Lipid Metabolism Disorders; Oxidative Stress
Keywords: Metabolism; Lipid oxidation; micronutrient cocktail supplementation; physical inactivity; glucose intolerance; oxidative stress
MeSH Terms: conditions — Glucose Intolerance; Sedentary Behavior; Glucose Metabolism Disorders; Lipid Metabolism Disorders | interventions — Docosahexaenoic Acids; Vitamin E; Selenium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Experimental): Intervention: Reduction in daily steps up to 2000-3000 steps per day and no structured physical activity + High dose ingestion of fructose (3g/kg/day) glucose (0,5g/kg/day)in the last 10 days of the protocol No cocktail during the protocol
  Healthy male volunteers in the active range of population (10000 to 15000 steps per day) aged 20-45 years, 22 BMI 27 158 cm height 190 cm, Certified as healthy by a comprehensive clinical assessment.
  Interventions: Dietary Supplement: control diet
- Cocktail intervention (Experimental): Intervention: Reduction in daily steps up to 2000-3000 steps per day and no structured physical activity + High dose ingestion of fructose (3g/kg/day) glucose (0,5g/kg/day)in the last 10 days of the protocol + Micronutrient cocktail supplementation with 560,7 mg/ day of polyphenols (3 pills/day), 2,1 g/day of omega-3 fatty-acids (3 pills/day), 168 mg/day of vitamin E and 80µg/day of selenium (1 pill/day)
  Healthy male volunteers in the active range of population (10000 to 15000 steps per day) aged 20-45 years, 22 BMI 27 158 cm height 190 cm, Certified as healthy by a comprehensive clinical assessment.
  Interventions: Dietary Supplement: XXS-2A + Omega-3 + Vitamin E + Selenium

INTERVENTIONS:
Dietary Supplement: XXS-2A + Omega-3 + Vitamin E + Selenium — Micronutrient cocktail supplementation with 560,7 mg/ day of polyphenols (3 pills/day), 2,1 g/day of omega-3 fatty-acids (3 pills/day), 168 mg/day of vitamin E and 80µg/day of selenium (1 pill/day)
  Arms: Cocktail intervention
Dietary Supplement: control diet — habitual diet to be followed
  Arms: Control

SUMMARY:
This experiment consists on a 20-day reduction in daily step in free-living active individuals to induce physical inactivity. This will be used to test the efficacy of the anti-oxidant cocktail we aim to test as a new countermeasure in 2016 during the 60-d bed rest planed by ESA/CNES.

The objective of this study is to investigate whether the cocktail of natural antioxidants XXS-2A comprising vitamin E and coupled with omega-3 helps to prevent and / or reduce the glucose intolerance and improve oxidative defenses induced by 20 days of physical inactivity through daily step reduction

Although physical inactivity is reported to affect glucose tolerance within days of inactivity, we selected a period of 20 days for the effect of the cocktail to take place and assess secondary molecular mechanisms. The effect of this short period of inactivity on metabolism will moreover be boosted during the last 10 days by taking fructose, a sugar found in abundance in fruits, honey and juices, which is known to quickly trigger metabolic deregulation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects,
* Aged 20-45 years,
* No obesity or excessive thinness with BMI (weight Kg / height m2) between 22 and 27,
* Height (cm) between 158 and 190 cm,
* Certified as healthy by a comprehensive clinical assessment (detailed medical history and complete physical examination): in particular, free from any chronic disease or any acute infectious disease or ENT, neurological, orthopaedic, musculoskeletal and cardiovascular disorders,
* In the active range of population (10000 to 15000 steps/day)
* No contraindication to lidocaïne,
* No allergy to peanuts or soya,
* Non smokers or smoking less than 5 cigarettes/day,
* No alcohol, no drug dependence and no medical treatment,

Regulations

* Having given written informed consent prior to any procedure related to the study,
* Covered by Health Insurance System,
* Not under any administrative or legal supervision,
* Not under guardianship or trusteeship.

Exclusion Criteria:

* Any history or presence of clinically relevant cardiovascular, neurological or ENT, any chronic disease; any acute infectious disease,
* Obesity or excessive thinness,
* Not in the active range of population (<10000 steps/day),
* Ongoing medical treatment,
* Poor tolerance to blood sampling,
* Having given blood (more than 8ml/kg) in a period of 8 weeks or less before the start of the experiment,
* Subject with contraindication to lidocaïne,
* Special food diet, vegetarian or vegan or food supplementation,
* History of food allergy, especially allergy to peanuts or soya,
* A significant history of allergy,
* Positive reaction to any of the following tests: HVA IgM (hepatitis A), HBs antigen (hepatitis B), anti-HVC antibodies (hepatitis C), anti-HIV1+2 antibodies,
* History or presence of drug or alcohol abuse (alcohol consumption > 40 grams/day).

General conditions

* Subject who, in the judgment of the Investigator, is likely to be non-compliant during the study, or unable to cooperate because of a language problem or poor mental development,
* Subject in the exclusion period of a previous study according to applicable regulations,
* Subject who has received more than 4500 Euros within 12 months for being a research subject,
* Subject who cannot be contacted in case of emergency,
* Incarcerated persons,
* Subject under guardianship or trusteeship.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in Lipid oxidation | 20 days
  change in lipid oxidation as measured by indirect calorimetry during a 4h-OGTT

SECONDARY OUTCOMES:
Change in glucose concentration | 20 days
  Change in plasma glucose concentration during a 4h-OGTT
Change in insulin concentration | 20 days
  Change in plasma insulin concentration during a 4h-OGTT
Change in NEFA | 20 days
  Change in fasting plasma NEFA
Change in triglycerides | 20 days
  Change in fasting plasma triglycerides
de novo lipogenesis | 20 days
  incorporation of labelled fructose in VLDL-TG
Change in fructose oxidation | 20 days
  Change in 13C recovery in breath samples from ingested 1-13C fructose
Change in oxidative stress | 20 days
  Change in fasting reduced and oxidized glutathione
Change in fat-free mass | 20 days
  Change in fat-free mass as measured by DXA
muscle pathways involved in intertwined protein synthesis / insulin sensitivity | 4h for each day of test. 12h for all the protocol
  western blots with Vastes lateralis samples obtained from muscle biopsy

CONTACTS AND LOCATIONS:
Locations (1):
- Medes-Imps, Toulouse, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Adams GR, Caiozzo VJ, Baldwin KM. Skeletal muscle unweighting: spaceflight and ground-based models. J Appl Physiol (1985). 2003 Dec;95(6):2185-201. doi: 10.1152/japplphysiol.00346.2003. PMID 14600160
- [Background] Alibegovic AC, Hojbjerre L, Sonne MP, van Hall G, Stallknecht B, Dela F, Vaag A. Impact of 9 days of bed rest on hepatic and peripheral insulin action, insulin secretion, and whole-body lipolysis in healthy young male offspring of patients with type 2 diabetes. Diabetes. 2009 Dec;58(12):2749-56. doi: 10.2337/db09-0369. Epub 2009 Aug 31. PMID 19720789
- [Background] Alibegovic AC, Sonne MP, Hojbjerre L, Bork-Jensen J, Jacobsen S, Nilsson E, Faerch K, Hiscock N, Mortensen B, Friedrichsen M, Stallknecht B, Dela F, Vaag A. Insulin resistance induced by physical inactivity is associated with multiple transcriptional changes in skeletal muscle in young men. Am J Physiol Endocrinol Metab. 2010 Nov;299(5):E752-63. doi: 10.1152/ajpendo.00590.2009. Epub 2010 Aug 24. PMID 20739510
- [Background] Bakker GC, van Erk MJ, Pellis L, Wopereis S, Rubingh CM, Cnubben NH, Kooistra T, van Ommen B, Hendriks HF. An antiinflammatory dietary mix modulates inflammation and oxidative and metabolic stress in overweight men: a nutrigenomics approach. Am J Clin Nutr. 2010 Apr;91(4):1044-59. doi: 10.3945/ajcn.2009.28822. Epub 2010 Feb 24. PMID 20181810
- [Background] Bergouignan A, Momken I, Lefai E, Antoun E, Schoeller DA, Platat C, Chery I, Zahariev A, Vidal H, Gabert L, Normand S, Freyssenet D, Laville M, Simon C, Blanc S. Activity energy expenditure is a major determinant of dietary fat oxidation and trafficking, but the deleterious effect of detraining is more marked than the beneficial effect of training at current recommendations. Am J Clin Nutr. 2013 Sep;98(3):648-58. doi: 10.3945/ajcn.112.057075. Epub 2013 Jul 31. PMID 23902784
- [Background] Bergouignan A, Momken I, Schoeller DA, Normand S, Zahariev A, Lescure B, Simon C, Blanc S. Regulation of energy balance during long-term physical inactivity induced by bed rest with and without exercise training. J Clin Endocrinol Metab. 2010 Mar;95(3):1045-53. doi: 10.1210/jc.2009-1005. Epub 2010 Jan 8. PMID 20061436
- [Background] Bergouignan A, Rudwill F, Simon C, Blanc S. Physical inactivity as the culprit of metabolic inflexibility: evidence from bed-rest studies. J Appl Physiol (1985). 2011 Oct;111(4):1201-10. doi: 10.1152/japplphysiol.00698.2011. Epub 2011 Aug 11. PMID 21836047
- [Background] Bergouignan A, Trudel G, Simon C, Chopard A, Schoeller DA, Momken I, Votruba SB, Desage M, Burdge GC, Gauquelin-Koch G, Normand S, Blanc S. Physical inactivity differentially alters dietary oleate and palmitate trafficking. Diabetes. 2009 Feb;58(2):367-76. doi: 10.2337/db08-0263. Epub 2008 Nov 18. PMID 19017764
- [Background] Bienso RS, Ringholm S, Kiilerich K, Aachmann-Andersen NJ, Krogh-Madsen R, Guerra B, Plomgaard P, van Hall G, Treebak JT, Saltin B, Lundby C, Calbet JA, Pilegaard H, Wojtaszewski JF. GLUT4 and glycogen synthase are key players in bed rest-induced insulin resistance. Diabetes. 2012 May;61(5):1090-9. doi: 10.2337/db11-0884. Epub 2012 Mar 8. PMID 22403297
- [Background] Biolo G, Agostini F, Simunic B, Sturma M, Torelli L, Preiser JC, Deby-Dupont G, Magni P, Strollo F, di Prampero P, Guarnieri G, Mekjavic IB, Pisot R, Narici MV. Positive energy balance is associated with accelerated muscle atrophy and increased erythrocyte glutathione turnover during 5 wk of bed rest. Am J Clin Nutr. 2008 Oct;88(4):950-8. doi: 10.1093/ajcn/88.4.950. PMID 18842781
- [Background] Blanc S, Normand S, Ritz P, Pachiaudi C, Vico L, Gharib C, Gauquelin-Koch G. Energy and water metabolism, body composition, and hormonal changes induced by 42 days of enforced inactivity and simulated weightlessness. J Clin Endocrinol Metab. 1998 Dec;83(12):4289-97. doi: 10.1210/jcem.83.12.5340. PMID 9851766
- [Background] Breen L, Stokes KA, Churchward-Venne TA, Moore DR, Baker SK, Smith K, Atherton PJ, Phillips SM. Two weeks of reduced activity decreases leg lean mass and induces "anabolic resistance" of myofibrillar protein synthesis in healthy elderly. J Clin Endocrinol Metab. 2013 Jun;98(6):2604-12. doi: 10.1210/jc.2013-1502. Epub 2013 Apr 15. PMID 23589526
- [Background] Buehlmeier J, Frings-Meuthen P, Remer T, Maser-Gluth C, Stehle P, Biolo G, Heer M. Alkaline salts to counteract bone resorption and protein wasting induced by high salt intake: results of a randomized controlled trial. J Clin Endocrinol Metab. 2012 Dec;97(12):4789-97. doi: 10.1210/jc.2012-2857. Epub 2012 Oct 1. PMID 23027921
- [Background] Cavanagh PR, Licata AA, Rice AJ. Exercise and pharmacological countermeasures for bone loss during long-duration space flight. Gravit Space Biol Bull. 2005 Jun;18(2):39-58. PMID 16038092
- [Background] Chavez JA, Knotts TA, Wang LP, Li G, Dobrowsky RT, Florant GL, Summers SA. A role for ceramide, but not diacylglycerol, in the antagonism of insulin signal transduction by saturated fatty acids. J Biol Chem. 2003 Mar 21;278(12):10297-303. doi: 10.1074/jbc.M212307200. Epub 2003 Jan 13. PMID 12525490
- [Background] Cree MG, Paddon-Jones D, Newcomer BR, Ronsen O, Aarsland A, Wolfe RR, Ferrando A. Twenty-eight-day bed rest with hypercortisolemia induces peripheral insulin resistance and increases intramuscular triglycerides. Metabolism. 2010 May;59(5):703-10. doi: 10.1016/j.metabol.2009.09.014. Epub 2009 Nov 17. PMID 19919871
- [Background] Fitts RH, Riley DR, Widrick JJ. Functional and structural adaptations of skeletal muscle to microgravity. J Exp Biol. 2001 Sep;204(Pt 18):3201-8. doi: 10.1242/jeb.204.18.3201. PMID 11581335
- [Background] Gwag T, Park K, Park J, Lee JH, Nikawa T, Choi I. Celastrol overcomes HSP72 gene silencing-mediated muscle atrophy and induces myofiber preservation. J Physiol Pharmacol. 2015 Apr;66(2):273-83. PMID 25903958
- [Background] Hargens AR, Bhattacharya R, Schneider SM. Space physiology VI: exercise, artificial gravity, and countermeasure development for prolonged space flight. Eur J Appl Physiol. 2013 Sep;113(9):2183-92. doi: 10.1007/s00421-012-2523-5. Epub 2012 Oct 19. PMID 23079865
- [Background] Heilbronn L, Smith SR, Ravussin E. Failure of fat cell proliferation, mitochondrial function and fat oxidation results in ectopic fat storage, insulin resistance and type II diabetes mellitus. Int J Obes Relat Metab Disord. 2004 Dec;28 Suppl 4:S12-21. doi: 10.1038/sj.ijo.0802853. PMID 15592481
- [Background] Hilder TL, Baer LA, Fuller PM, Fuller CA, Grindeland RE, Wade CE, Graves LM. Insulin-independent pathways mediating glucose uptake in hindlimb-suspended skeletal muscle. J Appl Physiol (1985). 2005 Dec;99(6):2181-8. doi: 10.1152/japplphysiol.00743.2005. Epub 2005 Aug 11. PMID 16099889
- [Background] Hilder TL, Tou JC, Grindeland RE, Wade CE, Graves LM. Phosphorylation of insulin receptor substrate-1 serine 307 correlates with JNK activity in atrophic skeletal muscle. FEBS Lett. 2003 Oct 9;553(1-2):63-7. doi: 10.1016/s0014-5793(03)00972-4. PMID 14550547
- [Background] Hirasaka K, Maeda T, Ikeda C, Haruna M, Kohno S, Abe T, Ochi A, Mukai R, Oarada M, Eshima-Kondo S, Ohno A, Okumura Y, Terao J, Nikawa T. Isoflavones derived from soy beans prevent MuRF1-mediated muscle atrophy in C2C12 myotubes through SIRT1 activation. J Nutr Sci Vitaminol (Tokyo). 2013;59(4):317-24. doi: 10.3177/jnsv.59.317. PMID 24064732
- [Background] Hokayem M, Blond E, Vidal H, Lambert K, Meugnier E, Feillet-Coudray C, Coudray C, Pesenti S, Luyton C, Lambert-Porcheron S, Sauvinet V, Fedou C, Brun JF, Rieusset J, Bisbal C, Sultan A, Mercier J, Goudable J, Dupuy AM, Cristol JP, Laville M, Avignon A. Grape polyphenols prevent fructose-induced oxidative stress and insulin resistance in first-degree relatives of type 2 diabetic patients. Diabetes Care. 2013 Jun;36(6):1454-61. doi: 10.2337/dc12-1652. Epub 2012 Dec 28. PMID 23275372
- [Background] Itani SI, Ruderman NB, Schmieder F, Boden G. Lipid-induced insulin resistance in human muscle is associated with changes in diacylglycerol, protein kinase C, and IkappaB-alpha. Diabetes. 2002 Jul;51(7):2005-11. doi: 10.2337/diabetes.51.7.2005. PMID 12086926
- [Background] Kanazashi M, Tanaka M, Murakami S, Kondo H, Nagatomo F, Ishihara A, Roy RR, Fujino H. Amelioration of capillary regression and atrophy of the soleus muscle in hindlimb-unloaded rats by astaxanthin supplementation and intermittent loading. Exp Physiol. 2014 Aug;99(8):1065-77. doi: 10.1113/expphysiol.2014.079988. Epub 2014 Jun 6. PMID 24907028
- [Background] Kelley DE. Skeletal muscle triglycerides: an aspect of regional adiposity and insulin resistance. Ann N Y Acad Sci. 2002 Jun;967:135-45. PMID 12079843
- [Background] Kelley DE, Goodpaster BH, Storlien L. Muscle triglyceride and insulin resistance. Annu Rev Nutr. 2002;22:325-46. doi: 10.1146/annurev.nutr.22.010402.102912. Epub 2002 Jan 4. PMID 12055349
- [Background] Knudsen SH, Hansen LS, Pedersen M, Dejgaard T, Hansen J, Hall GV, Thomsen C, Solomon TP, Pedersen BK, Krogh-Madsen R. Changes in insulin sensitivity precede changes in body composition during 14 days of step reduction combined with overfeeding in healthy young men. J Appl Physiol (1985). 2012 Jul;113(1):7-15. doi: 10.1152/japplphysiol.00189.2011. Epub 2012 May 3. PMID 22556394
- [Background] Krebs JM, Schneider VS, Evans H, Kuo MC, LeBlanc AD. Energy absorption, lean body mass, and total body fat changes during 5 weeks of continuous bed rest. Aviat Space Environ Med. 1990 Apr;61(4):314-8. PMID 2339966
- [Background] Krogh-Madsen R, Pedersen M, Solomon TP, Knudsen SH, Hansen LS, Karstoft K, Lehrskov-Schmidt L, Pedersen KK, Thomsen C, Holst JJ, Pedersen BK. Normal physical activity obliterates the deleterious effects of a high-caloric intake. J Appl Physiol (1985). 2014 Feb 1;116(3):231-9. doi: 10.1152/japplphysiol.00155.2013. Epub 2013 Nov 7. PMID 24201706
- [Background] Lee SM, Moore AD, Everett ME, Stenger MB, Platts SH. Aerobic exercise deconditioning and countermeasures during bed rest. Aviat Space Environ Med. 2010 Jan;81(1):52-63. doi: 10.3357/asem.2474.2010. PMID 20058738
- [Background] Machida S, Booth FW. Changes in signalling molecule levels in 10-day hindlimb immobilized rat muscles. Acta Physiol Scand. 2005 Feb;183(2):171-9. doi: 10.1111/j.1365-201X.2004.01395.x. PMID 15676058
- [Background] Margaritis I, Rousseau AS, Marini JF, Chopard A. Does antioxidant system adaptive response alleviate related oxidative damage with long term bed rest? Clin Biochem. 2009 Mar;42(4-5):371-9. doi: 10.1016/j.clinbiochem.2008.10.026. Epub 2008 Nov 24. PMID 19059391
- [Background] Mazzucco S, Agostini F, Biolo G. Inactivity-mediated insulin resistance is associated with upregulated pro-inflammatory fatty acids in human cell membranes. Clin Nutr. 2010 Jun;29(3):386-90. doi: 10.1016/j.clnu.2009.09.006. Epub 2009 Oct 28. PMID 19875212
- [Background] Momken I, Stevens L, Bergouignan A, Desplanches D, Rudwill F, Chery I, Zahariev A, Zahn S, Stein TP, Sebedio JL, Pujos-Guillot E, Falempin M, Simon C, Coxam V, Andrianjafiniony T, Gauquelin-Koch G, Picquet F, Blanc S. Resveratrol prevents the wasting disorders of mechanical unloading by acting as a physical exercise mimetic in the rat. FASEB J. 2011 Oct;25(10):3646-60. doi: 10.1096/fj.10-177295. Epub 2011 Jun 29. PMID 21715682
- [Background] Montani JP, Carroll JF, Dwyer TM, Antic V, Yang Z, Dulloo AG. Ectopic fat storage in heart, blood vessels and kidneys in the pathogenesis of cardiovascular diseases. Int J Obes Relat Metab Disord. 2004 Dec;28 Suppl 4:S58-65. doi: 10.1038/sj.ijo.0802858. PMID 15592488
- [Background] Morino K, Petersen KF, Shulman GI. Molecular mechanisms of insulin resistance in humans and their potential links with mitochondrial dysfunction. Diabetes. 2006 Dec;55 Suppl 2(Suppl 2):S9-S15. doi: 10.2337/db06-S002. PMID 17130651
- [Background] Ngo Sock ET, Le KA, Ith M, Kreis R, Boesch C, Tappy L. Effects of a short-term overfeeding with fructose or glucose in healthy young males. Br J Nutr. 2010 Apr;103(7):939-43. doi: 10.1017/S0007114509992819. Epub 2009 Nov 24. PMID 19930762
- [Background] Novelle MG, Wahl D, Dieguez C, Bernier M, de Cabo R. Resveratrol supplementation: Where are we now and where should we go? Ageing Res Rev. 2015 May;21:1-15. doi: 10.1016/j.arr.2015.01.002. Epub 2015 Jan 24. PMID 25625901
- [Background] O'Keefe MP, Perez FR, Sloniger JA, Tischler ME, Henriksen EJ. Enhanced insulin action on glucose transport and insulin signaling in 7-day unweighted rat soleus muscle. J Appl Physiol (1985). 2004 Jul;97(1):63-71. doi: 10.1152/japplphysiol.01361.2003. Epub 2004 Mar 5. PMID 15004002
- [Background] Ota N, Soga S, Haramizu S, Yokoi Y, Hase T, Murase T. Tea catechins prevent contractile dysfunction in unloaded murine soleus muscle: a pilot study. Nutrition. 2011 Sep;27(9):955-9. doi: 10.1016/j.nut.2010.10.008. Epub 2011 Jun 8. PMID 21641774
- [Background] Pavy-Le Traon A, Heer M, Narici MV, Rittweger J, Vernikos J. From space to Earth: advances in human physiology from 20 years of bed rest studies (1986-2006). Eur J Appl Physiol. 2007 Sep;101(2):143-94. doi: 10.1007/s00421-007-0474-z. Epub 2007 Jul 28. PMID 17661073
- [Background] Rector RS, Thyfault JP, Laye MJ, Morris RT, Borengasser SJ, Uptergrove GM, Chakravarthy MV, Booth FW, Ibdah JA. Cessation of daily exercise dramatically alters precursors of hepatic steatosis in Otsuka Long-Evans Tokushima Fatty (OLETF) rats. J Physiol. 2008 Sep 1;586(17):4241-9. doi: 10.1113/jphysiol.2008.156745. Epub 2008 Jul 10. PMID 18617560
- [Background] Ritz P, Acheson KJ, Gachon P, Vico L, Bernard JJ, Alexandre C, Beaufrere B. Energy and substrate metabolism during a 42-day bed-rest in a head-down tilt position in humans. Eur J Appl Physiol Occup Physiol. 1998 Sep;78(4):308-14. doi: 10.1007/s004210050425. PMID 9754970
- [Background] Ruderman NB, Saha AK, Vavvas D, Witters LA. Malonyl-CoA, fuel sensing, and insulin resistance. Am J Physiol. 1999 Jan;276(1):E1-E18. doi: 10.1152/ajpendo.1999.276.1.E1. PMID 9886945
- [Background] Rudwill F, Blanc S, Gauquelin-Koch G, Chouker A, Heer M, Simon C, Bergouignan A. Effects of different levels of physical inactivity on plasma visfatin in healthy normal-weight men. Appl Physiol Nutr Metab. 2013 Jun;38(6):689-93. doi: 10.1139/apnm-2012-0434. Epub 2013 Mar 8. PMID 23724888
- [Background] Sattar N, Scherbakova O, Ford I, O'Reilly DS, Stanley A, Forrest E, Macfarlane PW, Packard CJ, Cobbe SM, Shepherd J; west of Scotland coronary prevention study. Elevated alanine aminotransferase predicts new-onset type 2 diabetes independently of classical risk factors, metabolic syndrome, and C-reactive protein in the west of Scotland coronary prevention study. Diabetes. 2004 Nov;53(11):2855-60. doi: 10.2337/diabetes.53.11.2855. PMID 15504965
- [Background] Savage DB, Petersen KF, Shulman GI. Disordered lipid metabolism and the pathogenesis of insulin resistance. Physiol Rev. 2007 Apr;87(2):507-20. doi: 10.1152/physrev.00024.2006. PMID 17429039
- [Background] Servais S, Letexier D, Favier R, Duchamp C, Desplanches D. Prevention of unloading-induced atrophy by vitamin E supplementation: links between oxidative stress and soleus muscle proteolysis? Free Radic Biol Med. 2007 Mar 1;42(5):627-35. doi: 10.1016/j.freeradbiomed.2006.12.001. Epub 2006 Dec 15. PMID 17291986
- [Background] Sigaudo D, Fortrat JO, Allevard AM, Maillet A, Cottet-Emard JM, Vouillarmet A, Hughson RL, Gauquelin-Koch G, Gharib C. Changes in the sympathetic nervous system induced by 42 days of head-down bed rest. Am J Physiol. 1998 Jun;274(6):H1875-84. doi: 10.1152/ajpheart.1998.274.6.H1875. PMID 9841515
- [Background] Smith GI, Atherton P, Reeds DN, Mohammed BS, Rankin D, Rennie MJ, Mittendorfer B. Dietary omega-3 fatty acid supplementation increases the rate of muscle protein synthesis in older adults: a randomized controlled trial. Am J Clin Nutr. 2011 Feb;93(2):402-12. doi: 10.3945/ajcn.110.005611. Epub 2010 Dec 15. PMID 21159787
- [Background] Stein TP. Weight, muscle and bone loss during space flight: another perspective. Eur J Appl Physiol. 2013 Sep;113(9):2171-81. doi: 10.1007/s00421-012-2548-9. Epub 2012 Nov 29. PMID 23192310
- [Background] Stein TP, Leskiw MJ, Schluter MD, Hoyt RW, Lane HW, Gretebeck RE, LeBlanc AD. Energy expenditure and balance during spaceflight on the space shuttle. Am J Physiol. 1999 Jun;276(6 Pt 2):R1739-48. doi: 10.1152/ajpregu.1999.276.6.r1739. PMID 10362755
- [Background] Stein TP, Blanc S. Does protein supplementation prevent muscle disuse atrophy and loss of strength? Crit Rev Food Sci Nutr. 2011 Oct-Nov;51(9):828-34. doi: 10.1080/10408398.2010.482679. PMID 21888533
- [Background] Stein TP, Schluter MD, Galante AT, Soteropoulos P, Ramirez M, Bigbee A, Grindeland RE, Wade CE. Effect of hind limb muscle unloading on liver metabolism of rats. J Nutr Biochem. 2005 Jan;16(1):9-16. doi: 10.1016/j.jnutbio.2004.07.003. PMID 15629235
- [Background] Stein TP, Wade CE. Metabolic consequences of muscle disuse atrophy. J Nutr. 2005 Jul;135(7):1824S-1828S. doi: 10.1093/jn/135.7.1824S. PMID 15987873
- [Background] Stettler R, Ith M, Acheson KJ, Decombaz J, Boesch C, Tappy L, Binnert C. Interaction between dietary lipids and physical inactivity on insulin sensitivity and on intramyocellular lipids in healthy men. Diabetes Care. 2005 Jun;28(6):1404-9. doi: 10.2337/diacare.28.6.1404. PMID 15920059
- [Background] Tappy L, Le KA, Tran C, Paquot N. Fructose and metabolic diseases: new findings, new questions. Nutrition. 2010 Nov-Dec;26(11-12):1044-9. doi: 10.1016/j.nut.2010.02.014. Epub 2010 May 14. PMID 20471804
- [Background] Trudel G, Payne M, Madler B, Ramachandran N, Lecompte M, Wade C, Biolo G, Blanc S, Hughson R, Bear L, Uhthoff HK. Bone marrow fat accumulation after 60 days of bed rest persisted 1 year after activities were resumed along with hemopoietic stimulation: the Women International Space Simulation for Exploration study. J Appl Physiol (1985). 2009 Aug;107(2):540-8. doi: 10.1152/japplphysiol.91530.2008. Epub 2009 May 28. PMID 19478189
- [Background] Unger RH. Minireview: weapons of lean body mass destruction: the role of ectopic lipids in the metabolic syndrome. Endocrinology. 2003 Dec;144(12):5159-65. doi: 10.1210/en.2003-0870. Epub 2003 Sep 4. PMID 12960011
- [Background] van der Zijl NJ, Goossens GH, Moors CC, van Raalte DH, Muskiet MH, Pouwels PJ, Blaak EE, Diamant M. Ectopic fat storage in the pancreas, liver, and abdominal fat depots: impact on beta-cell function in individuals with impaired glucose metabolism. J Clin Endocrinol Metab. 2011 Feb;96(2):459-67. doi: 10.1210/jc.2010-1722. Epub 2010 Nov 17. PMID 21084401
- [Background] Vitadello M, Germinario E, Ravara B, Libera LD, Danieli-Betto D, Gorza L. Curcumin counteracts loss of force and atrophy of hindlimb unloaded rat soleus by hampering neuronal nitric oxide synthase untethering from sarcolemma. J Physiol. 2014 Jun 15;592(12):2637-52. doi: 10.1113/jphysiol.2013.268672. Epub 2014 Apr 7. PMID 24710058
- [Background] Zwart SR, Hargens AR, Smith SM. The ratio of animal protein intake to potassium intake is a predictor of bone resorption in space flight analogues and in ambulatory subjects. Am J Clin Nutr. 2004 Oct;80(4):1058-65. doi: 10.1093/ajcn/80.4.1058. PMID 15447920
- [Background] Zwart SR, Pierson D, Mehta S, Gonda S, Smith SM. Capacity of omega-3 fatty acids or eicosapentaenoic acid to counteract weightlessness-induced bone loss by inhibiting NF-kappaB activation: from cells to bed rest to astronauts. J Bone Miner Res. 2010 May;25(5):1049-57. doi: 10.1359/jbmr.091041. PMID 19874203
- [Derived] Damiot A, Demangel R, Noone J, Chery I, Zahariev A, Normand S, Brioche T, Crampes F, de Glisezinski I, Lefai E, Bareille MP, Chopard A, Drai J, Collin-Chavagnac D, Heer M, Gauquelin-Koch G, Prost M, Simon P, Py G, Blanc S, Simon C, Bergouignan A, O'Gorman DJ. A nutrient cocktail prevents lipid metabolism alterations induced by 20 days of daily steps reduction and fructose overfeeding: result from a randomized study. J Appl Physiol (1985). 2019 Jan 1;126(1):88-101. doi: 10.1152/japplphysiol.00018.2018. Epub 2018 Oct 4. PMID 30284519